CLINICAL TRIAL: NCT05899959
Title: Remote Cardiac Monitoring by the Corsano CardioWatch 287-2 Evaluation Study
Acronym: RECAMO
Status: Completed | Type: Observational
Sponsor: Corsano Health B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: RECAMO
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Rhythm; Disorder; Palpitations; Hypertension; Hypotension
Keywords: wristband; wearable; blood pressure; ekg; atrial fibrillation; hypertension; comparison
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Hypertension; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients receiving an EKG holter: patients receiving an EKG holter at the outpatient clinic for 24-48 hours of remote monitoring
  Interventions: Device: Corsano CardioWatch 287-2
- Patients receiving an automatic blood pressure cuff: patients receiving an automatic blood pressure cuff at the outpatient clinic for 24 hours of remote monitoring
  Interventions: Device: Corsano CardioWatch 287-2

INTERVENTIONS:
Device: Corsano CardioWatch 287-2 — Patients receive either an EKG holter or an automatic blood pressure cuff, as prescribed by their cardiologist. The readings from these devices (atrial fibrillation detection and blood pressure) will be compared to the readings from the CardioWatch 287-2.

SUMMARY:
In this study, a wristband that monitors hearth rhythm and blood pressure is assessed in free living conditions.

Two groups of patients are being recruited: patients receiving an EKG holter and patients receiving an automatic blood pressure monitor. Patients wear the wristband for 28 days. During this time, the number of atrial fibrillation episodes detected by the wristband is being counted, which is to be compared with the number of episodes detected by the holter. Also, blood pressure is measured continuously, which is to be compared with daily blood pressure measurements using a conventional blood pressure cuff.

DETAILED DESCRIPTION:
Background of the study:

Wearables have the potential to monitor patients remotely. The Corsano CardioWatch 287-2 is such a medical device that can monitor atrial fibrillation and long-term blood pressure. The device has been validated using clinical trials in hospitals, but validation in the intended remote setting is lacking.

Objective of the study:

Primary objective: To compare the number of episodes of atrial fibrillation detected by the Corsano CardioWatch 287-2 during 28 days of use with the number of episodes of atrial fibrillation detected by conventional Holter monitoring during 48 hours of use (standard care).

Secondary objective: To assess the difference in blood pressure measurements obtained by the Corsano CardioWatch 287-2 and the conventional cuff blood pressure monitor over a period of 28 days; to assess the usability of the Corsano CardioWatch 287-2 from a patient perspective.

Study design:

Group A:

Conventional 24 hour EKG holter monitoring will be compared to 28 day continuous monitoring by the Corsano CardioWatch 287-2 to assess whether the percentage of patients in whom atrial fibrillation is detected will increase. Detection of atrial fibrillation with the Corsano CardioWatch 287-2 is done by optical photoplethysmography (PPG), after which atrial fibrillation is confirmed with a 30-second ECG measurement.

Additionally, conventional cuff blood pressure will be compared to blood pressure measured by the Corsano CardioWatch 287-2 to validate free-living blood pressure monitoring. Patients will measure their blood pressure daily with a cuff blood pressure measurement device. The measurements at day 7, 14, 21 will be used to reinforce the Corsano blood pressure algorithm. The remaining measurements will be used to compare the blood pressure with the values measured by the Corsano CardioWatch 287-2 to assess accuracy.

Group B:

Conventional automatic cuff blood pressure measurement will be compared with the Corsano CardioWatch 287-2 for 24-48 hours. The automatic cuff blood pressure monitor will take a blood pressure reading every 30 minutes. Each reading will be compared with the Corsano CardioWatch 287-2 reading.

Study population:

Patients receiving a 24 hour EKG holter or an ambulant blood pressure device after visiting the cardiologist's outpatient clinic.

Primary study parameters/outcome of the study:

Absolute percentage increase of patients in whom at least one event of atrial fibrillation is detected by the Corsano CardioWatch 287-2 during 28 days of monitoring, compared to a conventional EKG holter during 24-48 hours of monitoring.

Secundary study parameters/outcome of the study (if applicable):

1. Mean blood pressure difference and its SD between blood pressure measured by the Corsano CardioWatch 287-2 and blood pressure measured by a conventional oscillometric blood pressure cuff.
2. Usability of the Corsano CardioWatch 287-2 in a remote care setting as determined by a questionnaire.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

At the cardiologist's office, Group A and B patients receive 3 blood pressure measurements. These are performed by a nurse. Group A will take daily blood pressure readings of themselves at home. If atrial fibrillation is detected by the wristband, Group A patients will be asked to take an ECG. Finally, Group A patients will be asked once to complete a questionnaire. Group B only has to wear the wristband for 24 to 48 hours as an additional burden in addition to the aforementioned initial measurements.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old;
* able to provide consent;
* receiving EKG holter or automatic blood pressure cuff for home monitoring per doctor prescription

Exclusion Criteria:

* Unable to wear the Corsano CardioWatch 287 due to reasons such as allergic reactions, wounds, amputations etc.;
* Unable to receive blood pressure measurements per cuff due to lymphedema, amputation, dialysis shunt, wounds, etc.;
* Pregnant women;
* Breastfeading women;
* Upper arm circumference not within the cuff range (22-42 cm)
* Unable or not willing to sign informed consent;
* Significant mental or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One group (A) receiving an EKG monitoring holter for the duration of 24 hours as part of standard care for atrial fibrillation screening. Besides, one group (B) receiving an automatic blood pressure cuff for the duration of 24 hours as part of standard care for blood pressure evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation detection rate | 28 days
  Absolute percentage increase of patients in whom at least one event of atrial fibrillation is detected by the Corsano CardioWatch 287-2 during 28 days of monitoring, compared to a conventional EKG holter during 24-48 hours of monitoring.
Blood pressure accuracy | 28 days (EKG holter group) or 1-2 days (Automatic blood pressure group)
  Mean systolic and diastolic blood pressure difference and its SD between blood pressure measured by the Corsano CardioWatch 287-2 and blood pressure measured by a conventional oscillometric blood pressure cuff.

SECONDARY OUTCOMES:
Blood pressure accuracy | 28 days (EKG holter group) or 1-2 days (Automatic blood pressure group)
  Bias and limits of agreement between systolic and diastolic blood pressure measured by the Corsano CardioWatch 287-2 and blood pressure measured by a conventional oscillometric blood pressure cuff.
Usability questionnaire | 28 days (EKG holter group) or 1-2 days (Automatic blood pressure group)
  Usability of the Corsano CardioWatch 287-2 in a remote care setting as assessed by a self-developed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Reinier de Graaf Gasthuis, Delft, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Vliet M, Aalberts JJJ, Hamelinck C, Hauer AD, Hoftijzer D, Monnink SHJ, Schipper JC, Constandse JC, Peters NS, Lip GYH, Steinhubl SR, Ronner E. Assessment of photoplethysmography-based blood pressure determinations during long-term and short-term remote cardiac monitoring: the RECAMO study. Eur Heart J Digit Health. 2025 Mar 27;6(4):763-771. doi: 10.1093/ehjdh/ztaf027. eCollection 2025 Jul. PMID 40703134
- [Derived] van Vliet M, Aalberts JJJ, Hamelinck C, Hauer AD, Hoftijzer D, Monnink SHJ, Schipper JC, Constandse JC, Peters NS, Lip GYH, Steinhubl SR, Ronner E. Ambulatory atrial fibrillation detection and quantification by wristworn AI device compared to standard holter monitoring. NPJ Digit Med. 2025 Mar 25;8(1):177. doi: 10.1038/s41746-025-01555-9. PMID 40133622